CLINICAL TRIAL: NCT02254551
Title: Phase II Trial of LDE225 (Sonidegib) Plus Bortezomib in Patients With Relapsed or Relapsed/Refractory Multiple Myeloma With a Dose-Finding Lead-In
Brief Title: Safety/Efficacy Study of LDE225 (Sonidegib) Plus Bortezomib in Patients With Relapsed or Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety lead-in data did not support continuation of study.
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MM 50
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2016-12

CONDITIONS: Multiple Myeloma
Keywords: relapsed multiple myeloma; refractory multiple myeloma; LDE225; Sonidegib; bortezomib; smoothened (SMO) inhibitors; Velcade
MeSH Terms: conditions — Multiple Myeloma | interventions — sonidegib; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDE225 Plus Bortezomib (Experimental): Lead-In Portion: The lead-in portion of this study will investigate the safety and tolerability, and determine the MTD of LDE225, in combination with bortezomib in this patient population.
  Expansion Portion: Eligible patients will receive LDE225 orally once daily for 21 days with the dose-level determined in the lead-in portion of the study. Eligible patients will also receive a standard regimen of bortezomib 1.3 mg/m2 on days 1, 4, 8, and 11 of each 21 day cycle.
  Maintenance Therapy: Patients who complete 16 cycles of therapy with stable disease or better will be eligible for single agent maintenance therapy of LDE225 at the MTD orally for up to 2 years or until progressive disease or unacceptable toxicity.
  Interventions: Drug: LDE225; Drug: Bortezomib

INTERVENTIONS:
Drug: LDE225 — Lead-In: LDE225 will be administered orally at three dose levels starting at 400mg. If acceptable tolerability is demonstrated, escalations may continue up to 800 mg. LDE225 will be administered orally as a single daily dose for 21 days in combination with a fixed dose of bortezomib to be given on Days 1, 4, 8, 11 of each 21 day cycle.
  Dose Expansion: LDE225 will be given as a single oral daily dose for 21 days at the MTD determined in the lead-in phase.
  Maintenance Therapy: Patients who complete 16 cycles of therapy with stable disease or better will be eligible for single agent maintenance therapy of LDE225 at the MTD orally for up to 2 years or until progressive disease or unacceptable toxicity.
  Other Names: Sonidegib
Drug: Bortezomib — In both the lead-in and dose expansion portions of the study, bortezomib, 1.3 mg/m2, will be administered by subcutaneous injection (SQ) on Days 1, 4, 8, 11 of each 21 day cycle.
  Other Names: Velcade

SUMMARY:
The purpose of the study is to determine whether the combination of LDE225 (sonidegib) plus bortezomib is safe and effective in the treatment of relapsed or relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
Although multiple myeloma (MM) is considered fatal, survival has dramatically improved with the introduction of more effective treatment options. Despite these advances, all patients eventually relapse and MM is generally considered incurable. LDE225 (Sonidegib) is an oral, investigational smoothened (SMO) inhibitor that has shown anti-tumor activity in certain cancers. Bortezomib is a highly active drug for the treatment of MM and has produced response rates in relapsed and/or refractory patients. This study will investigate the tolerability and feasibility of combining LDE225 with bortezomib in patients with bortezomib-sensitive relapsed or relapsed/refractory MM.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have measurable MM requiring systemic therapy defined as at least one of the following:

   * Serum M-protein ≥ 0.5 g/dL
   * Urine M-protein ≥ 200 mg/24 hrs
   * Serum free light chain assay: involved free light chain level ≥ 10 mg/dL provided the serum free light chain ratio is abnormal
2. Must have progressed during or after at least two previous treatment regimens. Patients who have received previous high dose therapy or autologous stem cell transplantation are eligible.
3. ECOG Performance Status score of 0-2.
4. Patients with adequate bone marrow, liver and renal function.
5. Patient is able to swallow and retain oral medication.
6. QTcF ≤450 msec for males and ≤ 470 msec for females on the screening ECG.
7. Female patients must not be of childbearing potential or must agree to use adequate contraceptive measures.
8. Male patients willing to use adequate contraceptive measures.
9. Willingness and ability to comply with study and follow-up procedures.
10. Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. Received any treatment for myeloma-directed treatment within 21 days. Localized radiation and dexamethasone must be completed within 7 days prior to study treatment
2. Refractory to bortezomib, defined as progression on or within 60 days of last bortezomib dose.
3. Received any investigational drug within 28 days or 5 half-lives (whichever is longer) prior to the first dose of LDE225. For other anti-neoplastic therapy (e.g., chemotherapy, targeted therapy or radiation), a minimum of 14 days between termination of the study drug and administration of LDE225 is required.
4. Patients who have previously been treated with systemic LDE225 or with other Hedgehog (Hh) pathway inhibitors.
5. Received major surgical procedures within 28 days of beginning study drug, or minor surgical procedures within 7 days. No waiting is required following port-a-cath placement.
6. Those who are pregnant or lactating.
7. Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study or potentially affect the interpretation of the study data.
8. Patients with > Grade 2 peripheral neuropathy (per NCI CTCAE V4.0) within 14 days prior to study enrollment.
9. Patients with a presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea Grade ≥2, and malabsorption syndrome).
10. Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as HMG CoA inhibitors (statins), clofibrate and gemfibrozil, and that cannot be discontinued at least 2 weeks prior to starting LDE225 treatment. If it is essential that the patient stays on a statin to control hyperlipidemia, only pravastatin may be used with extra caution.
11. Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment. Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on LDE225 treatment.
12. Receiving treatment with medications known to be moderate and strong inhibitors or inducers of CYP3A4 or CYP3A5, drugs that are BCRP substrates, or drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4 or CYP3A5 inhibitors should be discontinued at least 7 days prior to starting LDE225. Strong CYP3A4 or CYP3A5 inducers should be discontinued at least 2 weeks weeks weeks prior to starting treatment with LDE225.
13. Therapeutic doses of warfarin sodium or any other warfarin-derivative anticoagulants are not permitted since LDE225 is a competitive inhibitor of CYP2C9 based on the in vitro data. In this situation therapeutic anticoagulation may be accomplished using low molecular weight heparin (LMWH) or similar agents.
14. Those diagnosed with cardiac conditions currently or within last 6 months.
15. Those experiencing angina pectoris within 3 months.
16. Those who experienced acute myocardial infarction within 3 months.
17. Those with inadequately controlled hypertension defined as systolic blood pressure [SBP] > 180 mmHg or diastolic blood pressure (DBP) > 100 mmHg. Patients with values above these levels must have their blood pressure controlled with medication prior to starting treatment. Patients with a history of labile hypertension, or a history of poor compliance with an antihypertensive regimen are to be excluded.
18. Pregnant or lactating women, where pregnancy is confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
19. Patients who are not willing to apply highly effective contraception during the study and after the final dose of study treatment.
20. Sexually active males who are unwilling to use a condom during intercourse while taking drug and for 6 months after stopping investigational medications and agree not to father a child in this period.
21. Those with a serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
22. Those presenting with other active cancers, or history of treatment for invasive cancer within 3 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
23. Those with psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus G. Berdeja, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (5):
- United States (5):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Oncology Hematology Care, Cincinnati, Ohio
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Texas Transplant Institute/Methodist Healthcare, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The primary objective of this study was to investigate safety, tolerability and determine the maximum tolerated dose (MTD) of LDE225 to administer along with a fixed dose of bortezomib. Between March 2015 and September 2015, 7 patients were enrolled in the safety lead-in part of the study at 4 investigational sites in the U.S.
Pre-assignment Details: 7 patients received at least 1 cycle (21 days) of treatment on dose level 1.
Groups:
- LDE225 Plus Bortezomib: Safety Lead-In: To determine the maximum tolerated dose (MTD), LDE225 will be administered orally at three dose levels: 400mg, 600mg, and 800mg.
  Bortezomib will be administered by subcutaneous injection (SQ) at a fixed dose of 1.3 mg/m2 on days 1, 4, 8, and 11 of each 21 day cycle.
  Expansion: Patients will receive LDE225 orally once daily for 21 days at the MTD. Bortezomib will be administered SQ at a fixed dose of 1.3 mg/m2 on days 1, 4, 8, and 11 of each 21 day cycle.
  Maintenance Therapy: Patients who complete 16 cycles of therapy with stable disease or better will be eligible for single agent maintenance therapy of LDE225 at the MTD orally for up to 2 years or until progressive disease or unacceptable toxicity.
Period: Dose Escalation
Arm/Group | LDE225 Plus Bortezomib
Started | 7
Cohort 1: LDE225 400mg | 7 (1 patient was found to be refractory to bortezomib and deemed ineligible.)
Cohort 2: LDE225 600mg | 0
Cohort 3: LDE225 800mg | 0
Completed | 4 (Due to toxicity and lack of efficacy, no other dose levels were examined.)
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Dose-limiting toxicity | 2
Period: Expansion
Arm/Group | LDE225 Plus Bortezomib
Started | 0
Completed | 0
Not Completed | 0
Period: Maintenance
Arm/Group | LDE225 Plus Bortezomib
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LDE225 Plus Bortezomib
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 79 [52 to 84]
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5
  Black or African AMerican | 1
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of LDE225 Plus Bortezomib
Description: During the safety lead-in, a standard 3+3 dose escalation design was used to establish the MTD for LDE225 in combination with bortezomib. The MTD would be determined by the highest dose at which ≤1 of 6 patients experiences a dose-limiting toxicity (DLT) during one cycle (21 days) of therapy. If 2 of 6 patients within a dose level experienced a DLT, that dose level would be defined as exceeding MTD and no further dose escalation would occur. The previous dose level would be considered the MTD.
Time Frame: every 3 weeks up to 48 weeks
Measure: Number
Arm/Group | LDE225 Plus Bortezomib
Number analyzed (Participants) | 7
Value | NA — The MTD was not reached. Due to lack of efficacy and toxicity seen during dose level 1, additional dose levels were not examined and the study was terminated.

2. Primary Outcome: Time to Disease Progression
Description: Time to progression (TTP) is measured from Day 1 of study drug administration to disease progression using International Myeloma Working Group (IMWG) Uniform Response Criteria.
Time Frame: every 3 weeks up to 48 weeks, then every 3 months thereafter up to 3 years from initiation of study treatment.
Population: This outcome measure was to be assessed during the expansion phase of the study. The study closed early and did not proceed to this phase of the study. There is no data to report for this outcome measure.
Groups:
- LDE225 Plus Bortezomib: Safety Lead-In: LDE225 will be administered orally at three dose levels: 400mg, 600mg, and 800mg for 21 days.
  Bortezomib will be administered by subcutaneous injection (SQ) at a fixed dose of 1.3 mg/m2 on days 1, 4, 8, and 11 of each 21 day cycle.
  Expansion: Patients will receive LDE225 orally once daily for 21 days at the MTD. Bortezomib will be administered SQ at a fixed dose of 1.3 mg/m2 on days 1, 4, 8, and 11 of each 21 day cycle.
  Maintenance Therapy: Patients who complete 16 cycles of therapy with stable disease or better will be eligible for single agent maintenance therapy of LDE225 at the MTD orally for up to 2 years or until progressive disease or unacceptable toxicity.
Arm/Group | LDE225 Plus Bortezomib
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Response
Description: Number of patients with confirmed Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), Progressive Disease (PD) or Stable Disease (SD) according to International Myeloma Working Group (IMWG) Uniform Response Criteria. CR=5% or less plasma cells in bone marrow, disappearance of soft tissue plasmacytoma, negative immunofixation on serum and urine. VGPR=Serum and urine M-protein detectable by immunofixation but not by electrophoresis, disappearance of any soft tissue plasmacytomas that were present at baseline. PR= at least 50% reduction from baseline in serum M-protein and at least 90% reduction from baseline in 24hr urinary M-protein. PD=Increase of 25% or more from nadir in serum or urine proteins. SD= not meeting criteria for CR, VGPR, PR or PD.
Time Frame: Every 3 weeks up to 48 weeks
Population: Of 7 enrolled patients, 1 was deemed ineligible and was excluded from efficacy analyses. At a median follow-up of 6 weeks, 3 patients in Cohort 1 had progressive disease and 3 had stable disease. Study was terminated after reviewing data from this first lead-in cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | LDE225 Plus Bortezomib
Number analyzed (Participants) | 6
Participants
  Progressive Disease | 3
  Stable Disease | 3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected on Days 1 and 8 of every 21-day cycle for up to 48 weeks (plus 30 days for end of treatment visit).
Description: All patients who received at least one dose of LDE225 plus bortezomib.
Groups:
- Cohort 1: LDE225 400mg/m^2: Cohort 1 will receive LDE225 orally on a daily basis, at 400mg/m^2 every 21 days.
  Bortezomib will be administered by subcutaneous injection (SQ) at a fixed dose of 1.3 mg/m2 on days 1, 4, 8, and 11 of each 21 day cycle.
- Cohort 2: LDE225 600mg/m^2: Cohort 2 will receive LDE225 orally on a daily basis, at 600 mg every 21 days. Bortezomib will be administered by subcutaneous injection (SQ) at a fixed dose of 1.3 mg/m2 on days 1, 4, 8, and 11 of each 21 day cycle.
- Cohort 3: LDE225 800mg/m^2: Cohort 3 will receive LDE225 orally on a daily basis, at 800mg/m^2 every 21 days.
  Bortezomib will be administered by subcutaneous injection (SQ) at a fixed dose of 1.3 mg/m2 on days 1, 4, 8, and 11 of each 21 day cycle.
Arm/Group | Cohort 1: LDE225 400mg/m^2 | Cohort 2: LDE225 600mg/m^2 | Cohort 3: LDE225 800mg/m^2
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/7 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: LDE225 400mg/m^2 (N=7) | Cohort 2: LDE225 600mg/m^2 (N=0) | Cohort 3: LDE225 800mg/m^2 (N=0)
Viral Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events 4.03
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: LDE225 400mg/m^2 (N=7) | Cohort 2: LDE225 600mg/m^2 (N=0) | Cohort 3: LDE225 800mg/m^2 (N=0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Increased creatinine (Investigations) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Hyponatremia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Decreased creatinine clearance (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Investigations) | 3 (3) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination of study during dose-escalation did not support continuation of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.